CLINICAL TRIAL: NCT01626716
Title: Collaborative Care for Depressed Elderly in Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Hyeon Woo Yim, Professor, National Clinical Research Coordination Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A102065_2012_1
Record Dates: First submitted 2012-06-20; First posted 2012-06-25 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Depression; Elderly; Korean; Collaborative Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- case management (Experimental): patients who assigned to the intervention group will take 7 times phone calls from case manager
  Interventions: Other: care management
- control (No Intervention): usual care

INTERVENTIONS:
Other: care management — patients who assigned to the intervention group will take 7 times phone calls from case manager
  Arms: case management

SUMMARY:
Late-life depression is associated with physical limitations, greater functional impairment, increased utilization and cost of health care, and suicide. Collaborative care, linking primary and mental health specialty care, has been shown to be effective for the treatment of late-life depression in primary care settings in Western countries. The primary aim of this project is to implement a depression care management intervention, and examine its effectiveness on the depressive symptoms of older patients in Korean primary care settings. Based on chronic disease management theory and previous Collaborative care management studies in western countries, we propose to test a Depression Care Management intervention,which includes care manager to support a primary care physician of depression in their old patients. Care manager'd role are monitoring the progress of treatment, supporting patient's adherence, educating patients/ family and facilitate communication between providers. Also psychiatrists provide consultation and supervision of care managers. Using a randomized controlled design, we will examine whether the Depression care management is an effective treatment for patients with late life depression in rural Korea. The primary outcome would be the improvement of depressive symptoms of patients in primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* 60 year or older
* diagnosed depression based on DSM-IV criteria

Exclusion Criteria:

* impairment of hearing
* dementia
* other psychiatric disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reduced depression symptoms | 3 months
  HAMD (Hamilton Depression Ratind Scale) Difference HAMD score between the intervention and control group from baseline to 3 month follow-up

SECONDARY OUTCOMES:
Depression response and remissionhealth related quality of life | 3months and 6months
  HAMD (Hamilton Depression Ratind Scale) Depression response is defined by improvement 50% or more HAMD scores from baseline to each follow-up periods.
  Depression remission is defined by 7 or less of HAMD score at each follow-up periods
Reduced suicide ideation | 3 months and 6 months
  SSI (Beck's suicide ieation scale) Difference total SSI scores Between the two groups from baseline to each follow-up periods
Improvement of Quality of life | 3 months and 6 months
  EQ5D Difference EQ5D scores Between the two groups from baseline to each follow-up periods

CONTACTS AND LOCATIONS:
Locations (1):
- Chungju community health care center, Chungju, ChoongBuk, South Korea